CLINICAL TRIAL: NCT04929236
Title: Multicenter, Prospective, Double-Blinded, Parallel Group, Randomized Phase III Study to Evaluate Safety and Efficacy of Different PANZYGA Dose Regimens in Pediatric Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) Patients
Brief Title: Study to Evaluate Safety and Efficacy of Different PANZYGA Dose Regimens in Pediatric Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NGAM-11
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Chronic Inflammatory Demyelinating Polyneuropathy
MeSH Terms: interventions — Panzyga

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panzyga High Dose (Experimental): 2.0g/kg of PANZYGA administered intravenously every four weeks over a period of sixteen weeks for a total of five treatment dosages.
  Interventions: Drug: Panzyga
- Panzyga Low Dose (Experimental): 1.0g/kg of PANZYGA administered intravenously every four weeks over a period of sixteen weeks for a total of five treatment dosages.
  Interventions: Drug: Panzyga

INTERVENTIONS:
Drug: Panzyga — PANZYGA is a human immunoglobin solution with 10% protein content for intravenous (IV) administration.

SUMMARY:
Safety and Efficacy of Different PANZYGA Dose Regimens in Pediatric Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) Patients

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥2 years and ≤17 years.
2. Patients with a diagnosis of CIDP based on European Academy of Neurology/Peripheral Nerve Society (EANPNS) 2021 guidelone [1]
3. Clinical history of functional impairment due to CIDP, corresponding to an mRS score ≥2, but ≤5.
4. Voluntarily given written informed consent (provided by patient's parent or legal guardian) and assent (provided by the patient, if age appropriate per Independent Ethics Committee [IEC]/Institutional Research Board [IRB] requirements).

Exclusion Criteria:

1. Patients with previously diagnosed CIDP who lack any CIDP symptoms.
2. Patients with a known history of inherited neuropathy or a family history of inherited neuropathy.
3. Patients who have previously failed immunoglobulin therapy for CIDP.
4. Patients who received immunoglobulin or plasma exchange (PEX) within eight weeks prior to the Baseline Visit (washout phase). However, if a patient has clinical evidence of confirmed CIDP relapse during the washout phase (consistent with an increase in mRS of ≥1), they are eligible for trial enrolment.
5. Patients with a history of deep vein thrombosis (DVT) in the past year, or pulmonary embolism ever.
6. Patients on unstable (change in prescribed dose within the last eight weeks) corticosteroids or rituximab use.
7. Patients with known or suspected hypersensitivity, anaphylaxis, or severe systemic response to immune-globulins, blood or plasma derived products, or any component of PANZYGA.
8. Female patients who are breastfeeding, pregnant, or planning to become pregnant, or are unwilling to use an effective birth control method while on the study (acceptable methods of birth control for this study include: intrauterine device [IUD], hormonal contraception, male or female condom, spermicide gel, diaphragm, sponge, or cervical cap).
9. Presence of medical history information or clinical symptoms suggestive of human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) infections.
10. Severe liver and/or kidney disease (alanine aminotransferase [ALT] > 3 × upper limit of normal [ULN]; aspartate aminotransferase [AST] > 3 × ULN; and/or creatinine levels >44 µmol/L for children ages 2-3 years, >62 µmol/L for children ages 4-10 years, and >89 µmol/L for children ages 11-17 years.
11. Presence of medical history information or clinical symptoms suggestive of immunoglobulin (IgA) deficiency and antibodies against IgA.
12. History of alcohol or drug abuse in the previous year, per Investigator's opinion.
13. Unable or unwilling to comply with the study protocol.
14. Receipt of any other investigational medicinal product (IMP) within three months before study entry or participating in another interventional clinical study. Prior participation in an observational or open-label study involving an approved product may be allowed but require prior consultation with the Medical Monitor to assess eligibilty.
15. Any other condition(s) that, in the Investigator's opinion, makes it undesirable for the patient to participate in the study or may interfere with protocol compliance.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in CIDP Baseline | Up to 24 weeks
  Evaluate the efficacy of two PANZYGA dose regimens in pediatric CIDP patients based on change in CIDP symptoms, measured by the Modified Rankin Score. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 6.

SECONDARY OUTCOMES:
CIDP Relapse | Up to 24 weeks
  Evaluate percentage of patients with CIDP relapse between 2 doses of Panzyga with relapse defined as increase in Modified Rankin score by ≥1 point from the baseline score related to CIDP. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 6.
Time to CIDP Relapse | Up to 24 weeks
  Time to CIDP relapse or withdrawal for any other reason with with relapse defined as increase in Modified Rankin Score score by ≥1 point from the baseline score. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 6.
Percentage of Patients With Good/Excellent Response | Up to 24 weeks
  The percentage of patients with good/excellent response, defined by a Modified Rankin Score score of 0 or 1 in each arm at Week 24. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 6.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Octapharma Research Site, Birmingham, Alabama
  - Octapharma Research Site, Orange, California
  - Octapharma Research Site, Louisville, Kentucky
  - Octapharma Research Site, Philadelphia, Pennsylvania
  - Octapharma Research Site, Houston, Texas
  - Octapharma Research Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No